CLINICAL TRIAL: NCT02118337
Title: A Phase 1/2, Open-label Study to Evaluate the Safety and Antitumor Activity of MEDI0680 (AMP-514) in Combination With Durvalumab Versus Nivolumab Monotherapy in Subjects With Select Advanced Malignancies
Brief Title: A Phase 1/2, Open-label Study to Evaluate the Safety and Antitumor Activity of MEDI0680 (AMP-514) in Combination With Durvalumab Versus Nivolumab Monotherapy in Participants With Select Advanced Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6020C00001
Record Dates: First submitted 2014-04-11; First posted 2014-04-21 (Estimated); Results first posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Select Advanced Malignancies; Kidney Cancer; Clear Cell Renal Cell Carcinoma
Keywords: select advanced malignancies,; kidney cancer,; clear cell renal cell carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — durvalumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- MEDI0680 0.1 mg/kg + Durvalumab 3 mg/kg (Experimental): Participants in dose-escalation phase will receive IV infusion of MEDI0680 0.1 mg/kg and durvalumab 3 mg/kg every 2 weeks (Q2W) for up to 12 months.
  Interventions: Biological: MEDI0680; Biological: Durvalumab
- MEDI0680 0.1 mg/kg + Durvalumab 10 mg (Experimental): Participants in dose-escalation phase will receive IV infusion of MEDI0680 0.1 mg/kg and durvalumab 10 mg/kg Q2W for up to 12 months.
  Interventions: Biological: MEDI0680; Biological: Durvalumab
- MEDI0680 0.5 mg/kg + Durvalumab 10 mg (Experimental): Participants in dose-escalation phase will receive IV infusion of MEDI0680 0.5 mg/kg and durvalumab 10 mg/kg Q2W for up to 12 months.
  Interventions: Biological: MEDI0680; Biological: Durvalumab
- MEDI0680 2.5 mg/kg + Durvalumab 10 mg (Experimental): Participants in dose-escalation phase will receive IV infusion of MEDI0680 2.5 mg/kg and durvalumab 10 mg/kg Q2W for up to 12 months.
  Interventions: Biological: MEDI0680; Biological: Durvalumab
- MEDI0680 10 mg/kg + Durvalumab 10 mg (Experimental): Participants in dose-escalation phase will receive IV infusion of MEDI0680 10 mg/kg and durvalumab 10 mg/kg Q2W for up to 12 months.
  Interventions: Biological: MEDI0680; Biological: Durvalumab
- MEDI0680 20 mg/kg + Durvalumab 10 mg (Experimental): Participants in dose-escalation phase will receive IV infusion of MEDI0680 20 mg/kg and durvalumab 10 mg/kg Q2W for up to 12 months.
  Interventions: Biological: MEDI0680; Biological: Durvalumab
- MEDI0680 20 mg/kg (Experimental): Participants in dose-expansion phase will receive IV infusion of MEDI0680 20 mg/kg Q2W until unacceptable toxicity, confirmed disease progression, development of other reason for treatment discontinuation, or for a maximum of 2 years, whichever occurred first.
  Interventions: Biological: MEDI0680
- MEDI0680 20 mg/kg + Durvalumab 750 mg (Experimental): Participants in dose-expansion phase will receive IV infusion of MEDI0680 20 mg/kg and durvalumab 750 mg/kg Q2W until unacceptable toxicity, confirmed disease progression, development of other reason for treatment discontinuation, or for a maximum of 2 years, whichever occurred first.
  Interventions: Biological: MEDI0680; Biological: Durvalumab
- Nivolumab 240 mg (Active Comparator): Participants in dose-expansion phase will receive IV infusion of nivolumab 240 mg Q2W until unacceptable toxicity, confirmed disease progression, development of other reason for treatment discontinuation, or for a maximum of 2 years, whichever occurred first.
  Interventions: Biological: Nivolumab

INTERVENTIONS:
Biological: MEDI0680 — Participants will receive IV infusion of MEDI0680 0.1 or 0.5 or 2.5 or 10 or 20 mg/kg Q2W in dose-escalation phase and 20 mg/kg Q2W in dose-expansion phase.
  Other Names: AMP-514
  Arms: MEDI0680 0.1 mg/kg + Durvalumab 10 mg; MEDI0680 0.1 mg/kg + Durvalumab 3 mg/kg; MEDI0680 0.5 mg/kg + Durvalumab 10 mg; MEDI0680 10 mg/kg + Durvalumab 10 mg; MEDI0680 2.5 mg/kg + Durvalumab 10 mg; MEDI0680 20 mg/kg; MEDI0680 20 mg/kg + Durvalumab 10 mg; MEDI0680 20 mg/kg + Durvalumab 750 mg
Biological: Durvalumab — Participants will receive IV infusion of durvalumab 3 and 10 mg Q2W in dose-escalation phase and 750 mg Q2W in dose-expansion phase.
  Arms: MEDI0680 0.1 mg/kg + Durvalumab 10 mg; MEDI0680 0.1 mg/kg + Durvalumab 3 mg/kg; MEDI0680 0.5 mg/kg + Durvalumab 10 mg; MEDI0680 10 mg/kg + Durvalumab 10 mg; MEDI0680 2.5 mg/kg + Durvalumab 10 mg; MEDI0680 20 mg/kg + Durvalumab 10 mg; MEDI0680 20 mg/kg + Durvalumab 750 mg
Biological: Nivolumab — Participants will receive IV infusion of nivolumab 240 mg Q2W in dose-expansion phase.
  Arms: Nivolumab 240 mg

SUMMARY:
To evaluate the Safety and Antitumor Activity of MEDI0680 (AMP-514) in Combination with Durvalumab versus Nivolumab Monotherapy in Participants with Select Advanced Malignancies.

DETAILED DESCRIPTION:
This is a multicenter, open-label, Phase 1/2 study to evaluate the safety, tolerability, PK, immunogenicity, and antitumor activity of MEDI0680 in combination with durvalumab or nivolumab monotherapy in adult immunotherapy-naïve participants with selected advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years or older
* Eastern Cooperative Oncology Group performance status of 0-1
* Adequate organ function
* At least 1 prior line of therapy

Exclusion Criteria:

* Concurrent enrollment in another clinical study, unless in follow-up period or it is an observational study
* Concurrent chemotherapy, immunotherapy, biologic, or hormonal therapy for cancer treatment
* Prior treatment with immunotherapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2014-05-19 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Chow, MD, Principal Investigator — University of Washington; Omid Hamid, MD, Principal Investigator — The Angeles Clinic; Jhanelle Gray, MD, Principal Investigator — Moffitt Cancer Center; Rachel Sanborn, MD, Principal Investigator — Providence Cancer Center; Mohamad Salkeni, MD, Principal Investigator — Mary Babb Randolph Cancer Center; Monika Joshi, MD, Principal Investigator — Penn State Hershey Cancer Institute; Robert Alter, MD, Principal Investigator — John Theurer Cancer Center; Raid Aljumaily, MD, Principal Investigator — Peggy Charles Stephenson Cancer Center; Jason Chesney, MD, Principal Investigator — Brown Cancer Center; Fernando Quevedo, MD, Principal Investigator — Mayo Clinic; Martin Voss, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Johanna Bendell, Principal Investigator — SCRI Development Innovations, LLC; Elizabeth Henry, Principal Investigator — Loyola Univ. Medical Center; Lionel Lewis, Principal Investigator — Dartmouth-Hitchcock Medical Center; Brian Rini, Principal Investigator — The Cleveland Clinic; Peter Van Veldhuizen, Principal Investigator — Menorah Medical Center tour
Locations (27):
- United States (13):
  - Research Site, Los Angeles, California
  - Research Site, Tampa, Florida
  - Research Site, Overland Park, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Rochester, Minnesota
  - Research Site, Hackensack, New Jersey
  - Research Site, New York, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Hershey, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Seattle, Washington
- Australia (2):
  - Research Site, East Bentleigh
  - Research Site, Frankston
- Canada (2):
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- France (5):
  - Research Site, Bordeaux
  - Research Site, Dijon
  - Research Site, Marseille
  - Research Site, Paris
  - Research Site, Villejuif
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Groningen
- United Kingdom (3):
  - Research Site, Cambridge
  - Research Site, Cardiff
  - Research Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Voss MH, Azad AA, Hansen AR, Gray JE, Welsh SJ, Song X, Kuziora M, Meinecke L, Blando J, Achour I, Wang Y, Walcott FL, Oosting SF. A Randomized Phase II Study of MEDI0680 in Combination with Durvalumab versus Nivolumab Monotherapy in Patients with Advanced or Metastatic Clear-cell Renal Cell Carcinoma. Clin Cancer Res. 2022 Jul 15;28(14):3032-3041. doi: 10.1158/1078-0432.CCR-21-4115. PMID 35507017
- See also: Redacted Protocol D6020C00001 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6020C00001&attachmentIdentifier=3deba787-5852-4d7a-8a42-17800345394c&fileName=protocol-d6020c00001-amendment-5-Redacted.pdf&versionIdentifier=
- See also: Redacted SAP D6020C00001 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6020C00001&attachmentIdentifier=307a8dab-459e-49c8-8bfc-2c88593dcd87&fileName=D6020C00001_SAP_-Feb2018_-_FINAL_-_V3.0_final.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study is conducted in Australia, Canada, Europe and the USA.
Groups:
- MEDI0680 0.1 mg/kg + Durvalumab 3 mg: Participants in dose-escalation phase received IV infusion of MEDI0680 0.1 mg/kg and durvalumab 3 mg/kg every 2 weeks (Q2W) for up to 12 months.
- MEDI0680 0.1 mg/kg + Durvalumab 10 mg: Participants in dose-escalation phase received IV infusion of MEDI0680 0.1 mg/kg and durvalumab 10 mg/kg Q2W for up to 12 months.
- MEDI0680 0.5 mg/kg + Durvalumab 10 mg: Participants in dose-escalation phase received IV infusion of MEDI0680 0.5 mg/kg and durvalumab 10 mg/kg Q2W for up to 12 months.
- MEDI0680 2.5 mg/kg + Durvalumab 10 mg: Participants in dose-escalation phase received IV infusion of MEDI0680 2.5 mg/kg and durvalumab 10 mg/kg Q2W for up to 12 months.
- MEDI0680 10 mg/kg + Durvalumab 10 mg: Participants in dose-escalation phase received IV infusion of MEDI0680 10 mg/kg and durvalumab 10 mg/kg Q2W for up to 12 months.
- MEDI0680 20 mg/kg + Durvalumab 10 mg: Participants in dose-escalation phase received IV infusion of MEDI0680 20 mg/kg and durvalumab 10 mg/kg Q2W for up to 12 months.
- MEDI0680 20 mg/kg: Participants in dose-expansion phase received IV infusion of MEDI0680 20 mg/kg Q2W until unacceptable toxicity, confirmed disease progression, development of other reason for treatment discontinuation, or for a maximum of 2 years, whichever occurred first.
- MEDI0680 20 mg/kg + Durvalumab 750 mg: Participants in dose-expansion phase received IV infusion of MEDI0680 20 mg/kg and durvalumab 750 mg/kg Q2W until unacceptable toxicity, confirmed disease progression, development of other reason for treatment discontinuation, or for a maximum of 2 years, whichever occurred first.
- Nivolumab 240 mg: Participants in dose-expansion phase received IV infusion of nivolumab 240 mg Q2W until unacceptable toxicity, confirmed disease progression, development of other reason for treatment discontinuation, or for a maximum of 2 years, whichever occurred first.
Period: Overall Study
Arm/Group | MEDI0680 0.1 mg/kg + Durvalumab 3 mg | MEDI0680 0.1 mg/kg + Durvalumab 10 mg | MEDI0680 0.5 mg/kg + Durvalumab 10 mg | MEDI0680 2.5 mg/kg + Durvalumab 10 mg | MEDI0680 10 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg | MEDI0680 20 mg/kg + Durvalumab 750 mg | Nivolumab 240 mg
Started | 4 | 5 | 3 | 3 | 9 | 6 | 4 | 42 | 21
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 5 | 3 | 3 | 9 | 6 | 4 | 42 | 21
Not completed — Other | 1 | 0 | 0 | 0 | 2 | 3 | 1 | 28 | 15
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 2 | 1 | 2 | 2 | 1 | 4 | 2
Not completed — Death | 2 | 2 | 1 | 2 | 5 | 1 | 2 | 9 | 4

BASELINE CHARACTERISTICS:
Population: As-treated population included those participants who received any study drug (MEDI0680, durvalumab, or nivolumab) and grouped according to actual treatment received.
Groups:
- MEDI0680 0.1 mg/kg + Durvalumab 3 mg: Participants in dose-escalation phase received IV infusion of MEDI0680 0.1 mg/kg and durvalumab 3 mg/kg Q2W for up to 12 months.
- Total: Total of all reporting groups
Arm/Group | MEDI0680 0.1 mg/kg + Durvalumab 3 mg | MEDI0680 0.1 mg/kg + Durvalumab 10 mg | MEDI0680 0.5 mg/kg + Durvalumab 10 mg | MEDI0680 2.5 mg/kg + Durvalumab 10 mg | MEDI0680 10 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg | MEDI0680 20 mg/kg + Durvalumab 750 mg | Nivolumab 240 mg | Total
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 9 | 6 | 4 | 42 | 21 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (12.6) | 67.4 (8.4) | 52.3 (17.9) | 62.3 (11.6) | 62.1 (11.0) | 69.5 (9.9) | 64.8 (14.2) | 61.0 (9.8) | 59.1 (10.5) | 61.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 1 | 1 | 5 | 2 | 1 | 9 | 6 | 29
  Male | 3 | 2 | 2 | 2 | 4 | 4 | 3 | 33 | 15 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 6
  Not Hispanic or Latino | 3 | 5 | 2 | 2 | 7 | 6 | 4 | 40 | 20 | 89
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
  White | 4 | 4 | 3 | 2 | 8 | 6 | 3 | 34 | 16 | 80
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 7 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs) in Dose-escalation Phase
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through 90 days post end of treatment (approximately 5 years 10 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI0680 0.1 mg/kg + Durvalumab 3 mg | MEDI0680 0.1 mg/kg + Durvalumab 10 mg | MEDI0680 0.5 mg/kg + Durvalumab 10 mg | MEDI0680 2.5 mg/kg + Durvalumab 10 mg | MEDI0680 10 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg + Durvalumab 10 mg
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 9 | 6
Participants
  Any TEAE | 4 | 5 | 3 | 3 | 9 | 6
  Any TESAE | 1 | 1 | 1 | 2 | 6 | 0

2. Primary Outcome: Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs in Dose-escalation Phase
Description: Number of participants in dose-escalation phase with abnormal clinical laboratory parameters reported as TEAEs are reported. Abnormal clinical laboratory parameters are defined as any abnormal finding during analysis of serum chemistry, hematology, coagulation, and urine.
Time Frame: Day 1 through 90 days post end of treatment (approximately 5 years 10 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI0680 0.1 mg/kg + Durvalumab 3 mg | MEDI0680 0.1 mg/kg + Durvalumab 10 mg | MEDI0680 0.5 mg/kg + Durvalumab 10 mg | MEDI0680 2.5 mg/kg + Durvalumab 10 mg | MEDI0680 10 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg + Durvalumab 10 mg
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 9 | 6
Participants
  Anaemia | 0 | 0 | 1 | 1 | 3 | 0
  Iron deficiency anaemia | 0 | 0 | 0 | 0 | 1 | 0
  Leukocytosis | 1 | 0 | 0 | 0 | 0 | 0
  Lymphopenia | 0 | 0 | 0 | 0 | 1 | 0
  Activated partial thromboplastin time prolonged | 0 | 0 | 0 | 0 | 0 | 1
  Blood fibrinogen decreased | 1 | 0 | 0 | 0 | 0 | 1
  International normalized ratio | 0 | 0 | 0 | 0 | 0 | 1
  Lymphocyte count decreased | 0 | 0 | 0 | 0 | 0 | 1
  Prothrombin time prolonged | 0 | 0 | 0 | 0 | 0 | 1
  White blood cell count decreased | 0 | 0 | 0 | 0 | 0 | 1
  Alanine aminotransferase increased | 0 | 0 | 0 | 0 | 1 | 0
  Amylase increased | 0 | 0 | 0 | 0 | 1 | 1
  Aspartate aminotransferase increased | 0 | 0 | 0 | 0 | 2 | 0
  Blood alkaline phosphatase increased | 1 | 0 | 1 | 0 | 1 | 0
  Blood creatinine increased | 0 | 0 | 0 | 0 | 2 | 1
  Blood phosphorus decreased | 1 | 0 | 0 | 0 | 0 | 0
  Blood urea increased | 0 | 0 | 0 | 0 | 1 | 0
  Gamma glutamyltransferase increased | 0 | 0 | 0 | 0 | 1 | 0
  Lipase increased | 1 | 0 | 1 | 0 | 1 | 0
  Hypercalcaemia | 0 | 0 | 0 | 0 | 1 | 1
  Hyperglycaemia | 0 | 0 | 0 | 0 | 1 | 0
  Hyperkalaemia | 0 | 0 | 0 | 0 | 1 | 0
  Hypermagnesaemia | 0 | 0 | 1 | 0 | 0 | 0
  Hyperuricaemia | 1 | 0 | 0 | 0 | 1 | 0
  Hypoalbuminaemia | 0 | 0 | 0 | 0 | 1 | 0
  Hypokalaemia | 0 | 0 | 0 | 0 | 2 | 0
  Hypomagnesaemia | 0 | 0 | 0 | 0 | 2 | 0
  Hyponatraemia | 0 | 0 | 0 | 0 | 2 | 1
  proteinuria | 0 | 0 | 0 | 0 | 1 | 0

3. Primary Outcome: Number of Participants With Abnormal Vital Signs and Physical Examinations Reported as TEAES in Dose-escalation Phase
Description: Number of participants in dose-escalation phase with abnormal vital signs reported as TEAEs are reported. Abnormal vital signs is defined as any abnormal finding in the vital sign parameters (blood pressure, heart rate, body temperature, and respiratory rate). Abnormal physical examination findings are defined as any abnormal finding in the following body systems: head and neck, respiratory, cardiovascular, gastrointestinal, urogenital, musculoskeletal, neurological, psychiatric, dermatological, hematologic/lymphatic, and endocrine systems, and weight.
Time Frame: Day 1 through 90 days post end of treatment (approximately 5 years 10 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI0680 0.1 mg/kg + Durvalumab 3 mg | MEDI0680 0.1 mg/kg + Durvalumab 10 mg | MEDI0680 0.5 mg/kg + Durvalumab 10 mg | MEDI0680 2.5 mg/kg + Durvalumab 10 mg | MEDI0680 10 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg + Durvalumab 10 mg
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 9 | 6
Participants
  Atrial fibrillation | 0 | 0 | 0 | 0 | 1 | 0
  Palpitations | 1 | 0 | 0 | 0 | 0 | 0
  Sinus tachycardia | 0 | 0 | 0 | 0 | 1 | 0
  Tachycardia | 0 | 0 | 0 | 0 | 0 | 1
  Pyrexia | 0 | 0 | 2 | 0 | 3 | 1
  Weight decreased | 0 | 0 | 0 | 0 | 1 | 1
  Hypertension | 1 | 0 | 0 | 0 | 1 | 1

4. Primary Outcome: Number of Participants With Abnormal Electrocardiograms (ECGs) Reported as TEAEs in Dose-escalation Phase
Description: Number of participants in dose-escalation phase with abnormal ECG parameters reported as TEAEs are reported.
Time Frame: Day 1 through 90 days post end of treatment (approximately 5 years 10 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI0680 0.1 mg/kg + Durvalumab 3 mg | MEDI0680 0.1 mg/kg + Durvalumab 10 mg | MEDI0680 0.5 mg/kg + Durvalumab 10 mg | MEDI0680 2.5 mg/kg + Durvalumab 10 mg | MEDI0680 10 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg + Durvalumab 10 mg
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 9 | 6
Participants
  Palpitations | 1 | 0 | 0 | 0 | 0 | 0
  Atrial fibrillation | 0 | 0 | 0 | 0 | 1 | 0
  Sinus tachycardia | 0 | 0 | 0 | 0 | 1 | 0
  Pericardial effusion | 0 | 0 | 0 | 0 | 1 | 0
  Tachycardia | 0 | 0 | 0 | 0 | 0 | 1

5. Primary Outcome: Objective Response Rate (ORR) Based on Investigator-assessed Response Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) in Dose-expansion Phase
Description: The ORR is defined as best overall response of confirmed complete response (CR) or confirmed partial response (PR) based on RECIST v1.1. The CR is defined as disappearance of all target and non-target lesions and no new lesions. The PR is defined as >= 30% decrease in the sum of diameters of target lesions (compared to baseline) and no new non-target lesion. A confirmed CR or PR is defined as 2 CRs or 2 PRs that were separated by at least 4 weeks with no evidence of progression in-between.
Time Frame: From baseline (Day -42 to Day -1) through disease progression or end of treatment (approximately 5 years 10 months)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MEDI0680 20 mg/kg | MEDI0680 20 mg/kg + Durvalumab 750 mg | Nivolumab 240 mg
Number analyzed (Participants) | 4 | 42 | 21
Percentage of participants | 0 [0 to 60.2] | 16.7 [7.0 to 31.4] | 23.8 [8.2 to 47.2]
Statistical Analysis 1: Comparison: MEDI0680 20 mg/kg vs Nivolumab 240 mg; Test type: Superiority; p = 0.5494, Fisher Exact; Rate difference = -23.8, 95% CI 2-sided [-72.8 to 31.1]
Statistical Analysis 2: Comparison: MEDI0680 20 mg/kg + Durvalumab 750 mg vs Nivolumab 240 mg; Test type: Superiority; p = 0.5130, Fisher Exact; Rate difference = -7.1, 95% CI 2-sided [-33.6 to 20.0]

6. Secondary Outcome: Best Overall Response (BOR) Based on Investigator-assessed RECIST v1.1 in Dose-expansion Phase
Description: The BOR includes CR, PR, stable disease (SD), progressive disease (PD), and non-evaluable (NE) based on RECIST v1.1. The CR is defined as disappearance of all target and non-target lesions and no new lesions. The PR is defined as >= 30% decrease in the sum of diameters of target lesions (compared to baseline) and no new nontarget lesion. The PD is defined at least 20% decrease in the sum of diameters of target lesions (compared to baseline) and/or new lesion. The SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression. The NE is defined as either when no or only a subset of lesion measurements are made at an assessment.
Time Frame: From baseline (Day -42 to Day -1) through disease progression or end of treatment (approximately 5 years 10 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI0680 20 mg/kg | MEDI0680 20 mg/kg + Durvalumab 750 mg | Nivolumab 240 mg
Number analyzed (Participants) | 4 | 42 | 21
Participants
  CR | 0 | 2 | 0
  PR | 0 | 5 | 5
  SD | 3 | 17 | 8
  PD | 1 | 17 | 6
  NE | 0 | 1 | 2

7. Secondary Outcome: Disease Control Rate (DCR) Based on Investigator-assessed RECIST v1.1 in Dose-expansion Phase
Description: The DCR is defined as a BOR of confirmed CR, confirmed PR, or SD based on RECIST v1.1. A confirmed CR is defined as two CRs (disappearance of all target and non-target lesions and no new lesions) that were separated by at least 4 weeks with no evidence of progression in-between. A confirmed PR is defined as two PRs (>= 30% decrease in the sum of diameters of target lesions compared to baseline and no new non-target lesion) that were separated by at least 4 weeks with no evidence of progression in-between. The SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression. The DCR at >= 8 weeks and >=24 weeks are reported.
Time Frame: From baseline (Day -42 to Day -1) through disease progression or end of treatment (approximately 5 years 10 months)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MEDI0680 20 mg/kg | MEDI0680 20 mg/kg + Durvalumab 750 mg | Nivolumab 240 mg
Number analyzed (Participants) | 4 | 42 | 21
Percentage of participants
  DCR at >=8 weeks | 75.0 [19.4 to 99.4] | 57.1 [41.0 to 72.3] | 61.9 [38.4 to 81.9]
  DCR at >=24 weeks | 50.0 [6.8 to 93.2] | 38.1 [23.6 to 54.4] | 38.1 [18.1 to 61.6]

8. Secondary Outcome: Time to Response (TTR) Based on Investigator-assessed RECIST v1.1 in Dose-expansion Phase
Description: The TTR is defined as the time from the first dose of treatment until the first documentation of a subsequently confirmed OR (confirmed CR or confirmed PR) based on RECIST v1.1. A confirmed CR is defined as two CRs (disappearance of all target and non-target lesions and no new lesions) that were separated by at least 4 weeks with no evidence of progression in-between. A confirmed PR is defined as two PRs (>= 30% decrease in the sum of diameters of target lesions compared to baseline and no new non-target lesion) that were separated by at least 4 weeks with no evidence of progression in-between. The TTR was estimated using Kaplan-Meier method.
Time Frame: From baseline (Day -42 to Day -1) through disease progression or end of treatment (approximately 5 years 10 months)
Population: As-treated population included those participants who received any study drug (MEDI0680, durvalumab, or nivolumab) and grouped according to actual treatment received. The TTR was analyzed for those participants who achieved OR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MEDI0680 20 mg/kg | MEDI0680 20 mg/kg + Durvalumab 750 mg | Nivolumab 240 mg
Number analyzed (Participants) | 0 | 7 | 5
Months |  | 1.8 [1.7 to 9.1] | 1.8 [1.6 to 7.3]

9. Secondary Outcome: Duration of Response (DoR) Based on Investigator-assessed RECIST v1.1 in Dose-expansion Phase
Description: The DoR is defined as the duration from the first documentation of OR (confirmed CR or confirmed PR) to the first documented disease progression based on RECIST v1.1 or death due to any cause, whichever occurred first. A confirmed CR is defined as two CRs (disappearance of all target and non-target lesions and no new lesions) that were separated by at least 4 weeks with no evidence of progression in-between. A confirmed PR is defined as two PRs (>= 30% decrease in the sum of diameters of target lesions compared to baseline and no new non-target lesion) that were separated by at least 4 weeks with no evidence of progression in-between. The PD is defined at least 20% decrease in the sum of diameters of target lesions (compared to baseline) and/or new lesion. The DoR was estimated using Kaplan-Meier method.
Time Frame: From baseline (Day -42 to Day -1) through disease progression or end of treatment (approximately 5 years 10 months)
Population: As-treated population included those participants who received any study drug (MEDI0680, durvalumab, or nivolumab) and grouped according to actual treatment received. The DoR was analyzed for those participants who achieved OR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MEDI0680 20 mg/kg | MEDI0680 20 mg/kg + Durvalumab 750 mg | Nivolumab 240 mg
Number analyzed (Participants) | 0 | 7 | 5
Months |  | NA [12.9 to NA] — Median and upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | NA [4.4 to NA] — Median and upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis.

10. Secondary Outcome: Progression Free Survival (PFS) Based on Investigator-assessed RECIST v1.1 in Dose-expansion Phase
Description: The PFS is defined as the time from the start of study treatment until the first documentation of disease progression based on RECIST v1.1 or death due to any cause, whichever occurred first. The PFS was estimated using Kaplan-Meier method.
Time Frame: From baseline (Day -42 to Day -1) through disease progression or end of treatment (approximately 5 years 10 months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MEDI0680 20 mg/kg | MEDI0680 20 mg/kg + Durvalumab 750 mg | Nivolumab 240 mg
Number analyzed (Participants) | 4 | 42 | 21
Months | 5.5 [2.2 to 7.4] | 3.6 [2.0 to 5.5] | 3.6 [1.9 to 13.0]

11. Secondary Outcome: Overall Survival in Dose-expansion Phase
Description: The OS is defined as the time from the start of study treatment until death due to any cause. The OS was estimated using Kaplan-Meier method.
Time Frame: From baseline (Day -42 to Day -1) through disease progression or end of treatment (approximately 5 years 10 months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MEDI0680 20 mg/kg | MEDI0680 20 mg/kg + Durvalumab 750 mg | Nivolumab 240 mg
Number analyzed (Participants) | 4 | 42 | 21
Months | 19.9 [7.0 to 19.9] | NA [NA to NA] — Median and lower and upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | NA [12.0 to NA] — Median and upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis.

12. Secondary Outcome: BOR Based on Investigator-assessed Modified RECIST v1.1 in Dose-escalation Phase
Description: The BOR includes CR, PR, SD, PD, and NE per Modified RECIST v1.1. The CR is defined as disappearance of all target and non-target lesions and no new lesions. The PR is defined as >= 30% decrease in the sum of diameters of target lesions (compared to baseline) and no new nontarget lesion. The PD is defined at least 20% decrease in the sum of diameters of target lesions (compared to baseline) and/or new lesion. The SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression. The NE is defined as either when no or only a subset of lesion measurements are made at an assessment.
Time Frame: From baseline (Day -42 to Day -1) through disease progression or EOT (approximately 12 months for each participant)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI0680 0.1 mg/kg + Durvalumab 3 mg | MEDI0680 0.1 mg/kg + Durvalumab 10 mg | MEDI0680 0.5 mg/kg + Durvalumab 10 mg | MEDI0680 2.5 mg/kg + Durvalumab 10 mg | MEDI0680 10 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg + Durvalumab 10 mg
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 9 | 6
Participants
  CR | 0 | 0 | 0 | 0 | 1 | 0
  PR | 2 | 0 | 1 | 0 | 3 | 4
  SD | 1 | 1 | 0 | 1 | 2 | 1
  PD | 1 | 3 | 2 | 1 | 2 | 1
  NE | 0 | 1 | 0 | 1 | 1 | 0

13. Secondary Outcome: ORR Based on Investigator-assessed Modified RECIST v1.1 in Dose-escalation Phase
Description: The ORR is defined as best overall response of confirmed CR or confirmed PR based on modified RECIST v1.1. The CR is defined as disappearance of all target and non-target lesions and no new lesions. The PR is defined as >= 30% decrease in the sum of diameters of target lesions (compared to baseline) and no new non-target lesion. A confirmed CR or PR is defined as 2 CRs or 2 PRs that were separated by at least 4 weeks with no evidence of progression in-between.
Time Frame: From baseline (Day -42 to Day -1) through disease progression or EOT (approximately 12 months for each participant)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MEDI0680 0.1 mg/kg + Durvalumab 3 mg | MEDI0680 0.1 mg/kg + Durvalumab 10 mg | MEDI0680 0.5 mg/kg + Durvalumab 10 mg | MEDI0680 2.5 mg/kg + Durvalumab 10 mg | MEDI0680 10 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg + Durvalumab 10 mg
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 9 | 6
Percentage of participants | 50.0 [6.8 to 93.2] | 0 [0 to 52.2] | 33.3 [0.8 to 90.6] | 0 [0 to 70.8] | 44.4 [13.7 to 78.8] | 66.7 [22.3 to 95.7]

14. Secondary Outcome: DCR Based on Investigator-assessed Modified RECIST v1.1 in Dose-escalation Phase
Description: The DCR is defined as a BOR of confirmed CR, confirmed PR, or SD based on modified RECIST v1.1. A confirmed CR is defined as two CRs (disappearance of all target and non-target lesions and no new lesions) that were separated by at least 4 weeks with no evidence of progression in-between. A confirmed PR is defined as two PRs (>= 30% decrease in the sum of diameters of target lesions compared to baseline and no new non-target lesion) that were separated by at least 4 weeks with no evidence of progression in-between. The SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression. The DCR at >= 8 weeks and >=24 weeks are reported.
Time Frame: From baseline (Day -42 to Day -1) through disease progression or EOT (approximately 12 months for each participant)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MEDI0680 0.1 mg/kg + Durvalumab 3 mg | MEDI0680 0.1 mg/kg + Durvalumab 10 mg | MEDI0680 0.5 mg/kg + Durvalumab 10 mg | MEDI0680 2.5 mg/kg + Durvalumab 10 mg | MEDI0680 10 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg + Durvalumab 10 mg
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 9 | 6
Percentage of participants
  DCR at >= 8 weeks | 75.0 [19.4 to 99.4] | 20.0 [0.5 to 71.6] | 33.3 [0.8 to 90.6] | 33.3 [0.8 to 90.6] | 66.7 [29.9 to 92.5] | 83.3 [35.9 to 99.6]
  DCR at >= 24 weeks | 50.0 [6.8 to 93.2] | 0 [0 to 52.2] | 33.3 [0.8 to 90.6] | 0 [0 to 70.8] | 44.4 [13.7 to 78.8] | 83.3 [35.9 to 99.6]

15. Secondary Outcome: TTR Based on Investigator-assessed Modified RECIST v1.1 in Dose-escalation Phase
Description: The TTR is defined as the time from the first dose of treatment until the first documentation of a subsequently confirmed OR (confirmed CR or confirmed PR) based on modified RECIST v1.1. A confirmed CR is defined as two CRs (disappearance of all target and non-target lesions and no new lesions) that were separated by at least 4 weeks with no evidence of progression in-between. A confirmed PR is defined as two PRs (>= 30% decrease in the sum of diameters of target lesions compared to baseline and no new non-target lesion) that were separated by at least 4 weeks with no evidence of progression in-between. The TTR was estimated using Kaplan-Meier method.
Time Frame: From baseline (Day -42 to Day -1) through disease progression or EOT (approximately 12 months for each participant)
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MEDI0680 0.1 mg/kg + Durvalumab 3 mg | MEDI0680 0.1 mg/kg + Durvalumab 10 mg | MEDI0680 0.5 mg/kg + Durvalumab 10 mg | MEDI0680 2.5 mg/kg + Durvalumab 10 mg | MEDI0680 10 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg + Durvalumab 10 mg
Number analyzed (Participants) | 2 | 0 | 1 | 0 | 4 | 4
Months | 2.6 [1.6 to 3.5] |  | 3.4 [NA to NA] — Lower and upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. |  | 3.5 [1.6 to 3.5] | 3.2 [1.7 to 10.8]

16. Secondary Outcome: DoR Based on Investigator-assessed Modified RECIST v1.1 in Dose-escalation Phase
Description: The DoR is defined as the duration from the first documentation of OR (confirmed CR or confirmed PR) to the first documented disease progression based on modified RECIST v1.1 or death due to any cause, whichever occurred first. A confirmed CR is defined as two CRs (disappearance of all target and non-target lesions and no new lesions) that were separated by at least 4 weeks with no evidence of progression in-between. A confirmed PR is defined as two PRs (>= 30% decrease in the sum of diameters of target lesions compared to baseline and no new non-target lesion) that were separated by at least 4 weeks with no evidence of progression in-between. The PD is defined at least 20% decrease in the sum of diameters of target lesions (compared to baseline) and/or new lesion. The DoR was estimated using Kaplan-Meier method.
Time Frame: From baseline (Day -42 to Day -1) through disease progression or EOT (approximately 12 months for each participant)
Population: AAs-treated population included those participants who received any study drug (MEDI0680, durvalumab, or nivolumab) and grouped according to actual treatment received. The DoR was analyzed for those participants who achieved OR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MEDI0680 0.1 mg/kg + Durvalumab 3 mg | MEDI0680 0.1 mg/kg + Durvalumab 10 mg | MEDI0680 0.5 mg/kg + Durvalumab 10 mg | MEDI0680 2.5 mg/kg + Durvalumab 10 mg | MEDI0680 10 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg + Durvalumab 10 mg
Number analyzed (Participants) | 2 | 0 | 1 | 0 | 4 | 4
Months | 16.8 [NA to NA] — Lower and upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. |  | NA [NA to NA] — Median and lower and upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. |  | 7.4 [5.6 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | NA [5.6 to NA] — Median and upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis.

17. Secondary Outcome: PFS Based on Investigator-assessed Modified RECIST v1.1 in Dose-escalation Phase
Description: The PFS is defined as the time from the start of study treatment until the first documentation of disease progression based on modified RECIST v1.1 or death due to any cause, whichever occurred first. The PFS was estimated using Kaplan-Meier method.
Time Frame: From baseline (Day -42 to Day -1) through disease progression or EOT (approximately 12 months for each participant)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MEDI0680 0.1 mg/kg + Durvalumab 3 mg | MEDI0680 0.1 mg/kg + Durvalumab 10 mg | MEDI0680 0.5 mg/kg + Durvalumab 10 mg | MEDI0680 2.5 mg/kg + Durvalumab 10 mg | MEDI0680 10 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg + Durvalumab 10 mg
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 9 | 6
Months | 20.2 [1.6 to 20.2] | 1.7 [1.6 to 3.5] | 1.6 [1.6 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | 1.8 [1.5 to 3.4] | 7.0 [1.6 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | 23.4 [1.8 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis.

18. Secondary Outcome: OS in Dose-escalation Phase
Description: as for outcome 11
Time Frame: From baseline (Day -42 to Day -1) through disease progression or EOT (approximately 12 months for each participant)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MEDI0680 0.1 mg/kg + Durvalumab 3 mg | MEDI0680 0.1 mg/kg + Durvalumab 10 mg | MEDI0680 0.5 mg/kg + Durvalumab 10 mg | MEDI0680 2.5 mg/kg + Durvalumab 10 mg | MEDI0680 10 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg + Durvalumab 10 mg
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 9 | 6
Months | 16.3 [3.6 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | NA [4.2 to NA] — Median and upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | 14.7 [NA to NA] — Lower and upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | 7.9 [1.5 to 7.9] | 12.8 [3.1 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis. | NA [29.6 to NA] — Median and upper limit of 95% CI could not be derived due to insufficient events being observed at the time of the analysis.

19. Secondary Outcome: Number of Participants With TEAEs and TESAEs in Dose-expansion Phase
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through 90 days post end of treatment (approximately 5 years 10 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI0680 20 mg/kg | MEDI0680 20 mg/kg + Durvalumab 750 mg | Nivolumab 240 mg
Number analyzed (Participants) | 4 | 42 | 21
Participants
  Any TEAE | 4 | 42 | 20
  Any TESAE | 3 | 22 | 13

20. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs in Dose-expansion Phase
Description: Number of participants in dose-expansion phase with abnormal clinical laboratory parameters reported as TEAEs are reported. Abnormal clinical laboratory parameters defined as any abnormal finding during analysis of serum chemistry, hematology, coagulation, and urine.
Time Frame: Day 1 through 90 days post end of treatment (approximately 5 years 10 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI0680 20 mg/kg | MEDI0680 20 mg/kg + Durvalumab 750 mg | Nivolumab 240 mg
Number analyzed (Participants) | 4 | 42 | 21
Participants
  Anaemia | 1 | 6 | 5
  Neutropenia | 0 | 1 | 0
  Blood iron decreased | 0 | 0 | 1
  Lymphocyte count decreased | 0 | 0 | 1
  Neutrophil count decreased | 1 | 1 | 0
  Platelet count decreased | 0 | 0 | 1
  Platelet count increased | 0 | 0 | 1
  Prothrombin time prolonged | 0 | 0 | 1
  White blood cell count increased | 0 | 0 | 1
  Alanine aminotransferase increased | 1 | 1 | 3
  Amylase decreased | 0 | 0 | 1
  Amylase increased | 1 | 3 | 3
  Aspartate aminotransferase increased | 1 | 2 | 3
  Blood alkaline phosphatase increased | 0 | 0 | 1
  Blood bilirubin increased | 0 | 0 | 1
  Blood creatine increased | 1 | 1 | 0
  Blood creatine phosphokinase increased | 0 | 1 | 0
  Blood creatinine increased | 1 | 4 | 3
  Blood glucose increased | 0 | 0 | 1
  Blood triglycerides increased | 0 | 1 | 1
  C-reactive protein increased | 0 | 1 | 1
  Lipase increased | 1 | 4 | 2
  Transaminases increased | 0 | 1 | 0
  Hypercalcaemia | 0 | 6 | 2
  Hyperglycaemia | 0 | 1 | 0
  Hyperkalaemia | 0 | 2 | 2
  Hypertriglyceridaemia | 0 | 1 | 0
  Hypoalbuminaemia | 0 | 2 | 0
  Hypocalcaemia | 0 | 1 | 0
  Hypoglycaemia | 0 | 1 | 0
  Hypokalaemia | 0 | 5 | 2
  Hypomagnesaemia | 0 | 4 | 2
  Hyponatraemia | 1 | 3 | 1
  Hypophosphataemia | 0 | 1 | 3
  Urine abnormality | 0 | 1 | 0
  Blood thyroid stimulating hormone increased | 0 | 2 | 2
  Blood urine present | 0 | 0 | 1

21. Secondary Outcome: Number of Participants With Abnormal Vital Signs and Physical Examinations Reported as TEAEs in Dose-expansion Phase
Description: Number of participants in dose-expansion phase with abnormal vital signs reported as TEAEs are reported. Abnormal vital signs is defined as any abnormal finding in the vital sign parameters (blood pressure, heart rate, body temperature, and respiratory rate). Abnormal physical examination findings are defined as any abnormal finding in the following body systems: head and neck, respiratory, cardiovascular, gastrointestinal, urogenital, musculoskeletal, neurological, psychiatric, dermatological, hematologic/lymphatic, and endocrine systems, and weight.
Time Frame: Day 1 through 90 days post end of treatment (approximately 5 years 10 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI0680 20 mg/kg | MEDI0680 20 mg/kg + Durvalumab 750 mg | Nivolumab 240 mg
Number analyzed (Participants) | 4 | 42 | 21
Participants
  Atrial fibrillation | 0 | 2 | 1
  Tachycardia | 0 | 1 | 0
  Pyrexia | 2 | 9 | 2
  Weight decreased | 0 | 5 | 0
  Weight increased | 0 | 3 | 0
  Hypoxia | 0 | 1 | 1
  Hypertension | 1 | 5 | 0
  Hypotension | 1 | 2 | 1

22. Secondary Outcome: Number of Participants With Abnormal ECGs Reported as TEAEs in Dose-expansion Phase
Description: Number of participants in dose-expansion phase with abnormal ECG parameters reported as TEAEs are reported.
Time Frame: Day 1 through 90 days post end of treatment (approximately 5 years 10 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI0680 20 mg/kg | MEDI0680 20 mg/kg + Durvalumab 750 mg | Nivolumab 240 mg
Number analyzed (Participants) | 4 | 42 | 21
Participants
  Angina pectoris | 1 | 1 | 0
  Tachycardia | 0 | 1 | 0
  Atrial fibrillation | 0 | 2 | 1
  Cardiac failure congestive | 0 | 0 | 1

23. Secondary Outcome: Antitumor Activity of MEDI0680 and Durvalumab Versus Nivolumab Monotherapy in Immunotherapy-Naïve Participants With Advanced or Metastatic Clear-cell Renal Cell Carcinoma (ccRCC) Based on Blinded Independent Central Review (BICR) in Dose-expansion Phase
Time Frame: From baseline (Day -42 to Day -1) through disease progression or end of treatment (approximately 5 years 10 months)
Population: The study did not meet its primary endpoint of demonstrating superior antitumor effect of MEDI0680 in combination with durvalumab versus nivolumab monotherapy in immunotherapy-naïve participants with advanced or metastatic ccRCC as assessed by the investigator using RECIST v1.1. Therefore, the decision was made not to perform the BICR analysis for antitumor activity and hence data were not collected.
Arm/Group | MEDI0680 20 mg/kg | MEDI0680 20 mg/kg + Durvalumab 750 mg | Nivolumab 240 mg
Number analyzed (Participants) | 0 | 0 | 0

24. Secondary Outcome: Percent Change From Baseline in Tumor Size in Dose-escalation Phase (Based on Investigator-assessed Modified RECIST v1.1) and Dose-expansion Phase (Based on Investigator-assessed RECIST v1.1)
Time Frame: From baseline (Day -42 to Day -1) through disease progression or EOT (approximately 12 months for each participant for dose-escalation phase and approximately 5 years 10 months for dose-expansion phase)
Population: Per the Statistical Analysis Plan, the data for percent change from baseline in target lesion was to be presented using Spider plot analysis. Hence, numeric data were not collected for this outcome measure.
Arm/Group | MEDI0680 0.1 mg/kg + Durvalumab 3 mg | MEDI0680 0.1 mg/kg + Durvalumab 10 mg | MEDI0680 0.5 mg/kg + Durvalumab 10 mg | MEDI0680 2.5 mg/kg + Durvalumab 10 mg | MEDI0680 10 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg | MEDI0680 20 mg/kg + Durvalumab 750 mg | Nivolumab 240 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Serum Concentration of MEDI0680 in Dose-escalation and Dose-expansion Phases
Description: Serum concentration of MEDI0680 were assessed using parameters Cmin (pre-dose) and Cmax (end of infusion), where Cmin was trough concentration and Cmax was peak concentration.
Time Frame: Pre-dose and end of infusion on Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1
Population: As-treated population included those participants who received MEDI0680 and grouped according to actual treatment received. The "Number of participants Analyzed" denotes the number of participants who had quantifiable and calculable serum samples at the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | MEDI0680 0.1 mg/kg + Durvalumab 3 mg | MEDI0680 0.1 mg/kg + Durvalumab 10 mg | MEDI0680 0.5 mg/kg + Durvalumab 10 mg | MEDI0680 2.5 mg/kg + Durvalumab 10 mg | MEDI0680 10 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg | MEDI0680 20 mg/kg + Durvalumab 750 mg
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 9 | 6 | 4 | 40
μg/mL
  Cmin at Cycle1 Day1 | NA (NA) — The sample was not quantifiable; therefore, not calculable. | NA (NA) — The sample was not quantifiable; therefore, not calculable. | NA (NA) — The sample was not quantifiable; therefore, not calculable. | NA (NA) — The sample was not quantifiable; therefore, not calculable. | NA (NA) — The sample was not quantifiable; therefore, not calculable. | NA (NA) — The sample was not quantifiable; therefore, not calculable. | NA (NA) — The sample was not quantifiable; therefore, not calculable. | NA (NA) — The sample was not quantifiable; therefore, not calculable.
  Cmax at Cycle1 Day1: number analyzed (Participants) | 4 | 5 | 3 | 3 | 9 | 4 | 4 | 38
  Cmax at Cycle1 Day1 | 4.330 (26.18) | 3.877 (54.68) | 16.36 (26.46) | 69.28 (24.76) | 272.4 (24.62) | 529.9 (29.84) | 668.8 (21.04) | 135.9 (4007)
  Cmin at Cycle1 Day15: number analyzed (Participants) | 4 | 3 | 3 | 3 | 8 | 5 | 0 | 0
  Cmin at Cycle1 Day15 | 1.143 (22.70) | 0.9937 (35.93) | 4.428 (62.38) | 18.67 (12.88) | 46.87 (559.4) | 205.8 (24.56) |  |
  Cmax at Cycle1 Day15: number analyzed (Participants) | 4 | 3 | 3 | 3 | 8 | 5 | 0 | 0
  Cmax at Cycle1 Day15 | 5.420 (21.61) | 3.835 (25.30) | 20.52 (26.26) | 87.78 (20.69) | 348.1 (27.78) | 716.8 (26.72) |  |
  Cmin at Cycle2 Day1: number analyzed (Participants) | 4 | 4 | 3 | 3 | 7 | 6 | 4 | 36
  Cmin at Cycle2 Day1 | 1.645 (49.08) | 1.361 (38.07) | 7.879 (52.74) | 31.81 (4.480) | 155.7 (24.20) | 378.0 (17.95) | 308.6 (30.45) | 253.9 (52.11)
  Cmax at Cycle2 Day1: number analyzed (Participants) | 4 | 4 | 3 | 3 | 7 | 6 | 4 | 34
  Cmax at Cycle2 Day1 | 3.515 (145.9) | 3.688 (80.17) | 17.28 (56.32) | 92.07 (17.72) | 440.7 (28.18) | 860.8 (13.82) | 936.1 (24.91) | 586.6 (63.42)

26. Secondary Outcome: Serum Concentration of Durvalumab in Dose-escalation and Dose-expansion Phases
Description: Serum concentration of durvalumab were assessed using parameters Cmin (pre-dose) and Cmax (end of infusion), where Cmin was trough concentration and Cmax was peak concentration.
Time Frame: Pre-dose and end of infusion on Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1
Population: As-treated population included those participants who received durvalumab and grouped according to actual treatment received. The "Number of participants Analyzed" denotes the number of participants who had quantifiable and calculable serum samples at the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | MEDI0680 0.1 mg/kg + Durvalumab 3 mg | MEDI0680 0.1 mg/kg + Durvalumab 10 mg | MEDI0680 0.5 mg/kg + Durvalumab 10 mg | MEDI0680 2.5 mg/kg + Durvalumab 10 mg | MEDI0680 10 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg + Durvalumab 750 mg
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 9 | 6 | 41
μg/mL
  Cmin at Cycle1 Day1: number analyzed (Participants) | 4 | 5 | 3 | 3 | 9 | 6 | 38
  Cmin at Cycle1 Day1 | NA (NA) — The sample was not quantifiable; therefore, not calculable. | NA (NA) — The sample was not quantifiable; therefore, not calculable. | NA (NA) — The sample was not quantifiable; therefore, not calculable. | NA (NA) — The sample was not quantifiable; therefore, not calculable. | NA (NA) — The sample was not quantifiable; therefore, not calculable. | NA (NA) — The sample was not quantifiable; therefore, not calculable. | NA (NA) — The sample was not quantifiable; therefore, not calculable.
  Cmax at Cycle1 Day1 | 65.47 (10.02) | 216.1 (25.14) | 213.8 (9.943) | 188.0 (17.82) | 248.0 (27.20) | 253.9 (11.35) | 186.9 (33.42)
  Cmin at Cycle1 Day15: number analyzed (Participants) | 4 | 3 | 3 | 3 | 8 | 6 | 0
  Cmin at Cycle1 Day15 | 19.62 (16.49) | 63.02 (7.836) | 49.04 (80.97) | 86.10 (69.76) | 79.59 (63.46) | 70.31 (22.00) |
  Cmax at Cycle1 Day15: number analyzed (Participants) | 4 | 3 | 3 | 3 | 8 | 6 | 0
  Cmax at Cycle1 Day15 | 95.14 (12.79) | 245.8 (13.45) | 241.1 (30.90) | 225.0 (9.213) | 292.7 (33.84) | 321.8 (23.05) |
  Cmin at Cycle2 Day1: number analyzed (Participants) | 4 | 4 | 3 | 3 | 7 | 6 | 27
  Cmin at Cycle2 Day1 | 23.83 (14.35) | 83.76 (34.29) | 89.20 (56.00) | 136.3 (45.72) | 124.8 (55.78) | 142.5 (50.52) | 78.41 (55.62)
  Cmax at Cycle2 Day1: number analyzed (Participants) | 4 | 4 | 3 | 3 | 7 | 6 | 32
  Cmax at Cycle2 Day1 | 84.43 (17.13) | 280.9 (12.48) | 297.5 (42.41) | 267.0 (25.97) | 370.9 (42.57) | 342.3 (18.08) | 258.1 (28.36)

27. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADA) to MEDI0680 in Dose-escalation and Dose-expansion Phases
Description: Number of participants with positive ADAs to MEDI0680 are reported. Persistent positive is defined as positive at >= 2 post-baseline assessments (with >= 16 weeks between first and last positive) or positive at last post-baseline assessment. Transient positive is defined as negative at last post-baseline assessment and positive at only one post-baseline assessment or at >=2 post-baseline assessments (with <16 weeks between first and last positive).
Time Frame: Cycle 1 Day 1, Cycle 2 Day 1, Cycle 5 Day 1, Cycle 8 Day 1, Cycle 11 Day 1, 90 and 180 days post end of treatment (approximately 5 years and 10 months)
Population: As-treated population included those participants who received MEDI0680 and grouped according to actual treatment received. The "Number of participants Analyzed" denotes the number of participants evaluated for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI0680 0.1 mg/kg + Durvalumab 3 mg | MEDI0680 0.1 mg/kg + Durvalumab 10 mg | MEDI0680 0.5 mg/kg + Durvalumab 10 mg | MEDI0680 2.5 mg/kg + Durvalumab 10 mg | MEDI0680 10 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg | MEDI0680 20 mg/kg + Durvalumab 750 mg
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 8 | 6 | 4 | 39
Participants
  ADA positive post-baseline | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 2
  Persistent Positive | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Transient Positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

28. Secondary Outcome: Number of Participants With Positive ADA to Durvalumab in Dose-escalation and Dose-expansion Phases
Description: Number of participants with positive ADA to durvalumab are reported. Persistent positive is defined as positive at >= 2 post-baseline assessments (with >= 16 weeks between first and last positive) or positive at last post-baseline assessment. Transient positive is defined as negative at last post-baseline assessment and positive at only one post-baseline assessment or at >=2 post-baseline assessments (with <16 weeks between first and last positive).
Time Frame: as for outcome 27
Population: As-treated population included those participants who received durvalumab and grouped according to actual treatment received. The "Number of participants Analyzed" denotes the number of participants evaluated for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI0680 0.1 mg/kg + Durvalumab 3 mg | MEDI0680 0.1 mg/kg + Durvalumab 10 mg | MEDI0680 0.5 mg/kg + Durvalumab 10 mg | MEDI0680 2.5 mg/kg + Durvalumab 10 mg | MEDI0680 10 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg + Durvalumab 750 mg
Number analyzed (Participants) | 4 | 5 | 3 | 3 | 8 | 6 | 39
Participants
  ADA positive post-baseline | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Persistent Positive | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Transient Positive | 0 | 0 | 0 | 0 | 0 | 0 | 0

29. Secondary Outcome: ORR for Participants With Programmed Cell Death Ligand 1 (PD-L1) Status Positive and Negative in Dose-expansion Phase
Description: ORR for participants with PD-L1 status positive and negative are reported. The ORR is defined as best overall response of confirmed CR or confirmed PR based on RECIST v1.1. The CR is defined as disappearance of all target and non-target lesions and no new lesions. The PR is defined as >= 30% decrease in the sum of diameters of target lesions (compared to baseline) and no new non-target lesion. A confirmed CR or PR is defined as 2 CRs or 2 PRs that were separated by at least 4 weeks with no evidence of progression in-between.
Time Frame: From baseline (Day -42 to Day -1) through disease progression or end of treatment (approximately 5 years 10 months)
Population: As-treated population included those participants who received any study drug (MEDI0680, durvalumab, or nivolumab) and grouped according to actual treatment received. Participants with PD-L1 positive (> 1% tumor cell membrane or > 1% immune cell staining) and PD-L1 negative (<= 1% tumor cell membrane and <= 1% immune cell staining) were evaluated for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MEDI0680 20 mg/kg | MEDI0680 20 mg/kg + Durvalumab 750 mg | Nivolumab 240 mg
Number analyzed (Participants) | 4 | 42 | 21
Percentage of Participants
  Participants with PD-L1 positive: number analyzed (Participants) | 1 | 5 | 8
  Participants with PD-L1 positive | 0 [0 to 97.5] | 40.0 [5.3 to 85.3] | 37.5 [8.5 to 75.5]
  Participants with PD-L1 negative: number analyzed (Participants) | 3 | 37 | 13
  Participants with PD-L1 negative | 0 [0 to 70.8] | 13.5 [4.5 to 28.8] | 15.4 [1.9 to 45.4]

ADVERSE EVENTS:
Time Frame: Day 1 through 90 days post end of treatment (approximately 5 years 10 months)
Arm/Group | MEDI0680 0.1 mg/kg + Durvalumab 3 mg | MEDI0680 0.1 mg/kg + Durvalumab 10 mg | MEDI0680 0.5 mg/kg + Durvalumab 10 mg | MEDI0680 2.5 mg/kg + Durvalumab 10 mg | MEDI0680 10 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg + Durvalumab 10 mg | MEDI0680 20 mg/kg | MEDI0680 20 mg/kg + Durvalumab 750 mg | Nivolumab 240 mg
All-Cause Mortality (participants affected / at risk) | 2/4 | 2/5 | 1/3 | 2/3 | 5/9 | 1/6 | 2/4 | 9/42 | 4/21
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/5 | 1/3 | 2/3 | 6/9 | 0/6 | 3/4 | 22/42 | 13/21
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5 | 3/3 | 3/3 | 9/9 | 6/6 | 4/4 | 41/42 | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI0680 0.1 mg/kg + Durvalumab 3 mg (N=4) | MEDI0680 0.1 mg/kg + Durvalumab 10 mg (N=5) | MEDI0680 0.5 mg/kg + Durvalumab 10 mg (N=3) | MEDI0680 2.5 mg/kg + Durvalumab 10 mg (N=3) | MEDI0680 10 mg/kg + Durvalumab 10 mg (N=9) | MEDI0680 20 mg/kg + Durvalumab 10 mg (N=6) | MEDI0680 20 mg/kg (N=4) | MEDI0680 20 mg/kg + Durvalumab 750 mg (N=42) | Nivolumab 240 mg (N=21)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia of malignancy (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Colitis microscopic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic haemorrhage (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalitis autoimmune (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracranial mass (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI0680 0.1 mg/kg + Durvalumab 3 mg (N=4) | MEDI0680 0.1 mg/kg + Durvalumab 10 mg (N=5) | MEDI0680 0.5 mg/kg + Durvalumab 10 mg (N=3) | MEDI0680 2.5 mg/kg + Durvalumab 10 mg (N=3) | MEDI0680 10 mg/kg + Durvalumab 10 mg (N=9) | MEDI0680 20 mg/kg + Durvalumab 10 mg (N=6) | MEDI0680 20 mg/kg (N=4) | MEDI0680 20 mg/kg + Durvalumab 750 mg (N=42) | Nivolumab 240 mg (N=21)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 3 (5) | 0 (0) | 1 (2) | 6 (10) | 5 (29)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Hypercalcaemia of malignancy (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 2 (2)
Asthenopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Episcleritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Periorbital swelling (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 3 (4)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 12 (16) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 1 (3) | 2 (3) | 0 (0) | 0 (0) | 3 (12) | 5 (5) | 0 (0) | 15 (23) | 9 (14)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 3 (3)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (3) | 1 (1) | 1 (1) | 2 (3) | 5 (7) | 1 (3) | 3 (4) | 10 (13) | 7 (8)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 11 (15) | 6 (8)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (7) | 1 (1)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (2) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 2 (3) | 4 (4) | 19 (25) | 6 (7)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 2 (2) | 1 (1)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 0 (0) | 1 (1) | 5 (7) | 3 (4)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 8 (12) | 2 (3)
Secretion discharge (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Contrast media reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 3 (4) | 0 (0) | 3 (5) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 4 (5)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chemical burn of skin (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Cystitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Post procedural oedema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 1 (1) | 1 (3) | 3 (3)
Amylase decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (6) | 3 (8)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 2 (14) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 4 (5) | 3 (6)
Blood fibrinogen decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood iron decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood testosterone decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (3)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Eastern cooperative oncology group performance status worsened (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Electrocardiogram t wave abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical condition abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Influenza b virus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (2) | 0 (0) | 1 (3) | 0 (0) | 1 (5) | 0 (0) | 1 (2) | 4 (19) | 2 (12)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procalcitonin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Serum ferritin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tri-iodothyronine free abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 5 (7) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (4) | 0 (0) | 5 (5) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 1 (2)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 6 (9) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 2 (3) | 2 (5)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 5 (6) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (9) | 2 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 3 (4) | 1 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (8)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 10 (18) | 7 (12)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 10 (11) | 2 (2)
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 4 (5) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 6 (6) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (6) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 5 (6) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 6 (9) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 6 (7) | 4 (5)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (3) | 3 (3) | 4 (4)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 2 (3) | 0 (0) | 1 (2) | 6 (7) | 5 (7)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hyposmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 1 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 3 (3)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine abnormality (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Galactorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 1 (2) | 9 (17) | 8 (9)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 7 (9) | 8 (10)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 2 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 2 (2)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 7 (8) | 2 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 4 (7) | 2 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 4 (4)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 5 (10) | 0 (0) | 0 (0) | 7 (10) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 7 (9) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 4 (5)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Scar pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Xeroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 5 (7) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Vena cava embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises on going studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2017-03-29): https://cdn.clinicaltrials.gov/large-docs/37/NCT02118337/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT02118337/SAP_001.pdf